CLINICAL TRIAL: NCT06602349
Title: EFFICACY of USUAL MANAGEMENT of CHRONIC IDIOPATHIC ANO-PERINEAL PAIN by USING LOCAL ANESTHETIC INFILTRATION : a RANDOMIZED DOUBLE-BLIND SALINE-CONTROLLED TRIAL
Brief Title: EFFICACY of USUAL MANAGEMENT of CHRONIC IDIOPATHIC ANO-PERINEAL PAIN by USING LOCAL ANESTHETIC INFILTRATION
Acronym: EPHI-DACI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-001494-23
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Chronic Idiopathic Anopérineal Pain
Keywords: LIDOCAINE; posterior perineal block; randomized, double-blind; Salin solution; chronic idiopathic ano-perineal pain
MeSH Terms: interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental ARMS (Experimental): treated with lidocaine 10 mg/ml
  Interventions: Drug: Lidocaine 10 MG/ML
- placebo arm (Placebo Comparator): treated with placebo;salin solution
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lidocaine 10 MG/ML — administration of lidocaine in posterior perineal block infiltration
  Arms: experimental ARMS
Drug: Saline — administration of salin solution in posterior perineal block infiltration
  Arms: placebo arm

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of a posterior perineal block performed under neurostimulation at 1 month after local anesthetic infiltration in the treatment of chronic idiopathic ano-perineal pain.

The main questions aims to answer are :

1. The efficacy of a posterior perineal block performed under neurostimulation on pain 1 month after local anesthetic infiltration in the treatment of chronic idiopathic ano-perineal pain.
2. The rate of maintenance at 3 months of a positive response to the first infiltration.
3. The pain-free rate at 1 month after the first infiltration.
4. Evolution of quality of life and pain impact between inclusion and one month after the first infiltration.
5. Changes in anxiety and depressive disorders associated with pain between inclusion and one month after the first infiltration.
6. The evolution of symptoms related to central sensitization (both somatic and emotional) between inclusion and one month after the first infiltration.

Participants will :

* be managed with a posterior perineal block of lidocaine or saline solution under neurostimulation.
* complete a questionnaire on pain, anxiety and depression at inclusion and one month after injection of the research product (lidocaine or saline solution).

Researchers will compare between the two treatment arms (lidocaine versus saline solution) to see the rate of patients with a reduction of at least 3 points on a visual analog pain scale between inclusion and 1 month after the first injection.

DETAILED DESCRIPTION:
Chronic idiopathic ano-perineal pain (CICA) is defined as anoperineal pain involving the anal region that has been present for more than 3 months, and for which no cause has been identified on clinical examination or further investigations (MRI). The mechanisms underlying this pain are multiple, but involve the pudendal nerve in the majority of cases.

Therapeutic management of CDAD is based on 3 treatment strategies of progressively increasing aggressiveness: drug treatment, infiltrations and decompressive surgery.

Drug treatment is based on the empirical use of neuropathic pain medications with proven efficacy in other areas (shingles, diabetes, etc.). Patients are generally considered to be non-responders to drug treatment after failure (decrease in VAS scale < 3) of at least one antidepressant and one antiepileptic, whose dosages have been brought up to the maximum possible, or in whom a side effect has prevented the dose from being increased to its authorized maximum.

Therapeutic infiltrations most often involve the pudendal nerve (ITNP). Infiltration of the posterior branches of the sacrococcygeal roots is sometimes associated, to create a posterior perineal block (PPB). There is no consensus or recommendation on which molecules to use.

In most studies, a combination of local anesthetics and corticosteroids was used. However, Labat et al published the only randomized controlled trial comparing lidocaine infiltration of the pudendal nerve with or without methylprednisolone. Results were not significantly different (14% vs. 11%).

According to the literature, short-term pain relief up to 3 months was achieved in less than half of patients (11% to 39%) , and at 1 year, pain relief was still present in only around 10% (6.8% to 12.2%) of patients. The only recognized risk factor for failure appears to be the duration of pain (greater than 1 year). Other risk factors have been described in the literature, but only in one study and not in the others such as gender (male or female), age (over or under 70), duration of pain (over or under 1 year), and whether the pain is bilateral or not .

Currently, in our department, patients are treated with lidocaine BPP under neurostimulation. Given the poor results in terms of efficacy and the strong psychological component in chronic pain pathologies, investigators propose in this study to compare our usual management against placebo. Indeed, no type of infiltration has ever been compared to a placebo

-Main objective: evaluate the efficacy of BPP performed under neurostimulation on pain at 1 month after local anesthetic infiltration in the treatment of SCID.

Primary endpoint:

Comparison between the two treatment arms (lidocaine versus saline solution) of the rate of patients with a reduction of at least 3 points on a visual analog pain scale (VAS) between inclusion and 1 month after the first injection.

-Secondary objectives:

Compare between the two treatment arms:

1. 3-month maintenance rate of positive response to first infiltration.
2. Pain-free rate at 1 month after first infiltration.
3. Evolution of quality of life and pain impact between inclusion and one month after the first infiltration.
4. Change in anxiety and depressive disorders associated with pain between inclusion and one month after the first infiltration.
5. The evolution of symptoms related to central sensitization (both somatic and emotional) between inclusion and one month after the first infiltration.

At the end of the interventional phase, patients will be managed according to the department's usual procedures. Accepting patients will be included in a follow-up cohort for one year.

Secondary endpoints:

1. Maintenance of positive response at 3 months, defined as a reduction of at least 3 VAS points (compared with inclusion) 3 months after infiltration.
2. Percentage of patients with a VAS score equal to 0 at 1 month after the first infiltration.
3. Delta of the score on question 9 of the modified Concise Pain Questionnaire (CPQ) (French version of the Brief Pain Inventory) concerning the impact of pain .
4. Delta of scores A (anxiety dimension) and D (depression dimension) on the HAD scale
5. Delta of the score for part A of the French version of the CSI central sensitization score

Research procedures Placebo arm: Infiltration by injections of 6mL saline per injection site (left ischial-anal fossa, right ischial-anal fossa, coccyx).

Treatment arm: Infiltration by injections of 6mL lidocaine (10 mg/mL) per injection site (left ischio-anal fossa, right ischio-anal fossa, coccyx).

-Practical research procedure Pre-inclusion visit (D0-min 1 week) Eligible patients will be identified during the proctology consultation. They will be given an information note about the study and will have at least 1 week to think about it before the next consultation.

Inclusion visit and 1st infiltration (D0)

* Verification of inclusion/non-inclusion criteria
* Patient and physician sign consent form.
* Completion of scales and questionnaires (EVA, HAD, QCD, CSI).
* Randomization.
* Infiltration according to randomization arm.
* Collection of adverse events (AEs) and serious adverse events (SAEs) Visit 1 (D0+1month)
* Collection of adverse events (AEs) and serious adverse events (SAEs)
* Completion of scales and questionnaires (EVA, HAD, QCD, CSI). In the event of a negative response (decrease in VAS of less than 3 points), patients will be managed according to the department's routine.

Telephone call: patients with a positive response will be called two months later (i.e. 3 months after infiltration) for a telephone evaluation of VAS. In the event of a VAS increase of more than 2 points, a proctology consultation will be proposed.

Adverse events (AEs) and serious adverse events (SAEs) will also be recorded during the telephone call.

End-of-study visit:

* In the event of a negative response (decrease in VAS of less than 3 points), Visit 1 (1 month ±3 days) will correspond to the end-of-study visit;
* If the patient has a positive response, the end-of-study visit will correspond to the telephone visit (3 months +/- 1 week after infiltration).
* Number of patients This is a pilot study in which investigators plan to include 30 patients per arm, for a total of 60 patients.
* Statistical method The rate of successful patients at M1 between the two randomization arms will be analyzed using logistic regression, with treatment success or failure as the explanatory variable and randomization arm and duration of pain (stratification factor) as the explanatory variables.
* Provisional timetable Duration of inclusion period: 60 months Duration of participation of each subject: 3 months Total study duration: 63 months

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older,
* Express consent to participate in the study
* Affiliated or beneficiary of a social security plan
* Presenting chronic idiopathic ano-perineal pain
* MRI normal or without pathology explaining pain (Multidisciplinary consultation meeting reread if in doubt)
* Resistance to "standard" 1st-line medical treatment (level 1 or 2 analgesics and/or non-steroidal anti-inflammatory and/or local topicals)

Exclusion Criteria:

* Patient benefiting from a legal protection measure
* Pregnant or breast-feeding woman
* General and/or local infection (fistulous or cutaneous suppuration of anal margin) in progress
* Known neurological pathology that may explain pain
* Psychiatric pathology requiring medication
* Anticoagulants or haemostasis disorders
* Hypersensitivity to lidocaine hydrochloride or local anesthetics
* Recurrent porphyrias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2028-12-08 (Estimated); Study Completion 2029-03-08 (Estimated)

PRIMARY OUTCOMES:
Comparison between the two treatment arms (lidocaine versus saline) of the rate of patients with a reduction of at least 3 points on a visual analog pain scale (VAS) between inclusion and 1 month after the first injection. | 3 month
  Comparison between the two treatment arms (lidocaine versus saline) of the rate of patients with a reduction of at least 3 points on a visual analog pain scale (VAS)(lower value is 0 and means no pain, higher is 10 means the maximum of pain) between inclusion and 1 month after the first injection.
  The rate of successful patients at M1 between the two randomization arms will be analyzed using logistic regression, with treatment success or failure as the explanatory variable and randomization arm and duration of pain (stratification factor) as the explanatory variables.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe hospitalier Diaconesses Croix Saint Simon, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided
not yet decided